CLINICAL TRIAL: NCT04621019
Title: Evaluation of the Safety and the Efficacy of the of BTL-785F Device for Non-invasive Lipolysis and Circumference Reduction of the Abdomen
Brief Title: BTL-785F Device for Non-invasive Lipolysis and Circumference Reduction of the Abdomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785F_ABL
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Fat Burn
Keywords: lipolysis; circumference reduction; non-invasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-invasive lipolysis and circumference reduction of the abdomen (Experimental): The treatment administration phase consists of four (4) treatment visits, delivered at least 1 week apart. Follow-ups visits at 1 month and 3 months after the final treatment will be held.
  Interventions: Device: BTL-785F

INTERVENTIONS:
Device: BTL-785F — Treatment with study device.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-785F system equipped with BTL-785-1 applicator for non-invasive lipolysis (breakdown of fat) of the abdomen and reduction in circumference of the abdomen.

Safety measures will include documentation of adverse events (AE) during and after the procedures.

Follow-ups visits at 1 month and 3 months after the final treatment will be held.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for abdominal circumference reduction
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible fat deposits in the abdominal area as deemed appropriate by the Investigator (e.g. by pinch test or ultrasound fat thickness measurement)
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring and/or weight loss during study participation.
* No procedure for abdominal fat reduction (including cellulite treatment) in the last six months.
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting a significant change of weight in either direction during study participation.
* Willingness to comply with study instructions and to return to the clinic for required visits.

Exclusion Criteria:

* Bacterial or viral infection, acute inflammations
* Impaired immune system
* Isotretinoin use in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, etc.
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Sensitivity disorders in the treatment area
* Varicose veins, pronounced edemas
* Previous liposuction in the treatment area in the last six months
* Unstable weight within the last 6 months (change in weight ± 3%)
* Previous body contouring or cellulite treatments in the abdominal area in the last six months
* Any other disease or condition (e.g. hernia) at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Statistically significant reduction of abdominal fat thickness determined with ultrasound | 5 months
  To gather clinical evidence that BTL-785F system equipped with BTL-785-1 applicator is able to provide statistically significant reduction of at least 1,5 cm at the 3-months follow-up compared to baseline with a minimum response rate of 65% in both abdominal circumference and fat thickness.

SECONDARY OUTCOMES:
Evaluation of the safety of the BTL-785F device with BTL-785-1 applicator for non-invasive lipolysis and circumference reduction of the abdomen | 5 months
  At every treatment visit after the first, prior to the procedure, the participants will be assessed for adverse effects resulting from the previous treatment(s) with the BTL-785F device.
  Safety measures will include documentation of adverse events (AE) during and after the procedures.
Assessment of the participants' satisfaction from the therapy measured via standard questionnaire | 5 months
  Minimum 80% of treated subjects to report satisfaction (level satisfied and higher) with the therapy;

CONTACTS AND LOCATIONS:
Locations (2):
- Bulgaria (2):
  - Ambulatory for Individual Practice for Specialized Outpatient Medical Care in Dermatology and Venereology Dr. Ivelina Yordanova-Vasileva, Pleven
  - Dr. Lekova Derm Ltd., Sofia

IPD SHARING:
Plan to Share IPD: No